CLINICAL TRIAL: NCT01374620
Title: Phase I Study : Dose Escalation of Intravenous Weekly Paclitaxel in Association With Metronomic Administration of Cyclophosphamide
Brief Title: Weekly Paclitaxel and Cyclophosphamide in Metronomic Administration : Dose Escalation Study of Weekly Paclitaxel
Acronym: PAL-ANGI2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAL-ANGI2
Record Dates: First submitted 2011-06-14; First posted 2011-06-16 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Cancer
Keywords: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Paclitaxel; Cyclophosphamide; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paclitaxel Dose escalation (Experimental): A standard dose escalation strategy will be used including 3 to 6 patients at each dose level (Paclitaxel dose escalation + fixed dose of cyclophosphamide)
  + blood collection
  Interventions: Drug: Paclitaxel dose escalation; Drug: Cyclophosphamide; Biological: Blood collection
- Cohort extension (Experimental): An additional 10 patients will be treated at the recommended dose in order to confirm the recommended paclitaxel dose
  + blood collection
  Interventions: Drug: Paclitaxel; Drug: Cyclophosphamide; Biological: Blood collection

INTERVENTIONS:
Drug: Paclitaxel dose escalation — Paclitaxel will be administered intravenously over 60 minutes, at D1, D8 and D15, at a given dose.
  The Paclitaxel dose (mg/infusion) levels are as follows:
  * 40
  * 60
  * 70
  * 75
  * 80
  * 85
  * 90
  Other Names: Taxol
  Arms: Paclitaxel Dose escalation
Drug: Paclitaxel — Patients will be treated at the recommended dose in order to confirm the recommended paclitaxel dose in association with metronomic cyclophosphamide
  Other Names: Taxol
  Arms: Cohort extension
Drug: Cyclophosphamide — D1 to D28: 50 mg x 2/day/cycle
  1 cycle = 28 days
  Other Names: Endoxan
Biological: Blood collection — At D1, D8, D15 and D21 of cycle 1 and cycle 2:2 blood samples for the correlation between clinical response and biological parameters

SUMMARY:
The aim of the study is to determine the MTD of Paclitaxel in association with metronomic Cyclophosphamide.

DETAILED DESCRIPTION:
The aim of the study is to determine the MTD of Paclitaxel in association with metronomic Cyclophosphamide for cancer which present no therapeutic solution

ELIGIBILITY:
Inclusion Criteria:

* Patient with cancer histologically proved
* No other therapeutic proposal after discussion in multidisciplinary consultation
* Radiological evidence of the evolving nature of the disease
* Measurable disease with at least one measurable lesion according to the criteria RECIST 1.1
* At least 28 days since prior treatment(systemic treatment or major surgery)
* Patient who have recovered from any previous toxicity
* Man or woman de ≥ 18 years and ≤ 65 years
* Performance Status (ECOG) ≤ 2 within 7 days before inclusion
* Polynuclear neutrophils ≥ 1500/mm3, platelets ≥ 100 000/mm3, Hemoglobin ≥ 9 g/dl
* Serum Albumin ≥ 36 g/l and lymphocytes ≥ 700/mm3
* Total bilirubin and SGPT/ALT and SGOT/AST ≤ 3 ULN(≤ 5 ULN if liver metastases)
* Creatinine in normal ranges and Creatinine clairance > 60 ml/min (Cockroft formulae)
* Central venous access
* Negative pregnancy test for women who may be pregnant within 7 days before inclusion
* Effective contraceptive during the treatment period and up to 6 months after the end of treatment (for patients of both sexes during their reproductive and child-bearing age and their partners)
* Patient covered by government health insurance
* Informed consent signed by the patient before any specific study procedure

Exclusion Criteria:

* Prior treatment by Paclitaxel
* Oral treatment impossible
* Known dysphagia, malabsorption or maldigestion
* Pre-existing neuropathy clinically symptomatic
* Known leptomeningeal brain metastases
* Known allergy to Cremophor, to Paclitaxel or one of its excipients (especially polyoxyethylene castor oil), to Cyclophosphamide or one of its excipients (lactose, sucrose)
* Active and uncontrolled infection
* Acute urinary tract infection, pre-existing hemorrhagic cystitis
* Diabetes insipidus
* History or progressive psychiatric illness
* Persons under guardianship or detainees
* Unable for medical follow-up (geographic, social or mental reasons)
* Pregnant, or likely to be or breastfeeding women
* Absence of effective contraception for the duration of treatment and 6 months after completion of therapy (for patients of both sexes in childbearing or reproductive age and their partners)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-06; Primary Completion 2013-02 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Determination of the iv paclitaxel maximum tolerated dose and recommended dose in association with a fixed dose of oral cyclophosphamide | 28 days = cycle 1
  A DLT is defined below:
  Hematological toxicity:
  * Polunuclear neutrophils < 500/mm3 for more than 7 days
  * Febrile neutropenia (Polunuclear neutrophils < 1 000/mm3 and fever > or = 38.5°C) or documented infection
  * Thrombopenia (Platelets < 25 000/mm3)
  * Impossibility to administer D8 or D15 due to hematological critera
  Non-hematological toxicity:
  Any grade 3 or 4 toxicity related to study treatment, with the exception of fatigue and alopecia

SECONDARY OUTCOMES:
Description of the nature of adverse events | During the study treatment, an expected average of 2 months
  According to the NCI-CTCAE scale v4.0
Evaluation of objective response after 2 cycles | After 2 cycles = 2 months
  Objective response (complete response, partial response and stable disease) according to RECIST 1.1 criteria
Estimation of the free-progression median time | Until disease progression
  Time between the inclusion and the disease progression (clinical or radiological)
Calculation of the Growth Modulation Index (GMI) | Until disease progression
  Time to progression on study treatment and time to progression on prior treatment
Evaluation of the correlation between clinical response and biological parameters | Day 1, 8, 15, 21 of cycle 1 and cycle 2
  Biological parameters related to angiogenesis
Description of the severity of adverse events | During the study treatment, an expected average of 2 months
  According to the NCI-CTCAE scale v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas PENEL, MD, Principal Investigator — Centre Oscar Lambret
Locations (1):
- Centre Oscar Lambret, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pannier D, Adenis A, Bogart E, Dansin E, Clisant-Delaine S, Decoupigny E, Lesoin A, Amela E, Ducornet S, Meurant JP, Le Deley MC, Penel N. Once weekly paclitaxel associated with a fixed dose of oral metronomic cyclophosphamide: a dose-finding phase 1 trial. BMC Cancer. 2018 Jul 31;18(1):775. doi: 10.1186/s12885-018-4678-x. PMID 30064401